CLINICAL TRIAL: NCT06134076
Title: Impact of Fermented Pulses on Inflammation and the Gut Microbiota
Brief Title: Comparing Effects of Fermented and Unfermented Pulses and Gut Microbiota
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Darrell W. Cockburn, Ph.D., Assistant Professor, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: STUDY00023162; 58-3060-3-052 (Other Grant/Funding Number: USDA ARS)
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Fermented Food; Inflammation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: 2 week run-in period with no pulse consumption. Randomly assigned to order of receiving interventions. Blood sample, fecal sample, dietary recall. 2 week intervention 1. Blood sample, fecal sample, dietary recall. 2 week washout. 2 week intervention 2. Blood sample, fecal sample, dietary recall.
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will receive both interventions labeled only as 1 or 2. The study team assessing inflammation and microbiome will not know the identity of intervention 1 or 2. The preparer of the meals will also conduct dietary recall interviews with subjects and will know the identities of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Unfermented Chickpea (Experimental)
  Interventions: Other: Unfermented chickpea
- Fermented Chickpea (Experimental)
  Interventions: Other: Fermented chickpea

INTERVENTIONS:
Other: Unfermented chickpea — Frozen meals containing 100 g unfermented chickpeas
  Arms: Unfermented Chickpea
Other: Fermented chickpea — Frozen meals containing 100 g fermented chickpeas
  Arms: Fermented Chickpea

SUMMARY:
The goal of this clinical trial is to learn about the effects of consuming fermented pulses (certain types of legumes like chickpeas or lentils) in healthy people. The main questions it aims to answer are:

1. How does consuming the fermented foods impact the gut microbiome?
2. Does this interaction between the fermented foods and the gut microbiome affect inflammation?

Participants will be asked to consume two sets of prepared meals, one containing unfermented pulses, the other containing fermented pulses.

Researchers will compare the gut microbiome and inflammation between these two diets.

DETAILED DESCRIPTION:
The rationale for the research is that fermentation of pulses can reduce the concentration of compounds that suppress butyrate producing bacteria and butyrate production. This will in turn boost butyrate production during consumption of these fermented pulses relative to that in unfermented pulses. This in turn will lead to lower inflammation in people consuming fermented pulses. To best study this question the investigators will utilize a cross-over design trial where participants will consume daily meals containing either fermented or unfermented pulses (chickpeas), followed by a washout period and then a period of consuming the other type of pulse. The investigators hypothesize that those consuming the fermented pulses will experience a significant decrease in inflammatory markers driven by increased butyrate production by gut bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults

Exclusion Criteria:

* Taken antibiotics within the past month
* Taking any medication for the management of diabetes or obesity
* Are pregnant
* BMI > 24.9
* Allergies to pulses or any other meal components

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in inflammation levels from baseline and between interventions | At 2 weeks (baseline), 4 weeks (after first intervention), 8 weeks (after second intervention)
  Measured in blood (IL-1β, IL-6, IL-10, IL-12, IFN-γ, TNF-α) and in feces (NGAL, calprotectin)

SECONDARY OUTCOMES:
Change in fecal short chain fatty acids from baseline and between interventions | At 2 weeks (baseline), 4 weeks (after first intervention), 8 weeks (after second intervention)
  Measurement of acetate, propionate and butyrate in feces
Change in gut microbiome composition from baseline and between interventions | At 2 weeks (baseline), 4 weeks (after first intervention), 8 weeks (after second intervention)
  Measured by fecal 16S rRNA gene sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Cockburn, PhD, Principal Investigator — Penn State University

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers, only summarized data